CLINICAL TRIAL: NCT01643824
Title: A Phase II Study Using Hypofractionated Proton Beam Radiotherapy for Hepatocellular Carcinoma
Brief Title: Hypofractionated Proton Beam Radiotherapy for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-12-622
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Proton Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Beam Therapy (Experimental): * Prescription dose to PTV as according to the following dose escalation schema: Arml 1: 60 GyE /10 fx, 6GyE fraction dose, 5 days/week, for HCC free from the alimentary tract (i.e., stomach, duodenum, esophagus, small and large bowel) (more than 2cm from clinical target volume), TLV30 <40%, and/or RLV30 <30%) Arm 2: 50 GyE /10 fx, 5GyE fraction dose, 5 days/week, for HCC close to the alimentary tract (less than 2cm from clinical target volume) but not contact with the alimentary tract, TLV30<50% and RLV30<40% Arm 3: 35 GyE /10 fx, 4GyE fraction dose, 5 days/week, for HCC contact to the alimentary tract (contact with clinical target volume), TLV30<60%, and/or RLV30<50%
  * Dose prescription : 95% isodose volume of prescribed dose encompassed PTV
  Interventions: Radiation: Proton Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — - Prescription dose to PTV as according to the following dose escalation schema: Arml 1: 60 GyE /10 fx, 6GyE fraction dose, 5 days/week, for HCC free from the alimentary tract (i.e., stomach, duodenum, esophagus, small and large bowel) (more than 2cm from clinical target volume), TLV30 <40%, and/or RLV30 <30%) Arm 2: 50 GyE /10 fx, 5GyE fraction dose, 5 days/week, for HCC close to the alimentary tract (less than 2cm from clinical target volume) but not contact with the alimentary tract, TLV30<50% and RLV30<40% Arm 3: 35 GyE /10 fx, 4GyE fraction dose, 5 days/week, for HCC contact to the alimentary tract (contact with clinical target volume), TLV30<60%, and/or RLV30<50%
  - Dose prescription : 95% isodose volume of prescribed dose encompassed PTV
  Other Names: Radiotherapy

SUMMARY:
This phase II study is to evaluate the effectiveness of hypofractionated proton beam therapy (PBT) for HCC patients in hepatitis B endemic area.

DETAILED DESCRIPTION:
The primary endpoint is local progression free survival. The trial is a single arm phase II trial with the historical arm. The expected 3-year local progression free survival for patient with HCC patients treated with proton beam therapy would be 80%. With a power of 80% and a type I error level of 10%, evaluable 40 patients are required to reject that the null hypothesis that true 3-year local progression free survival rate is ≤65%. Considering the 10% unevaluable patients due to loss of follow up, a total 45 eligible patients for each arms will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed as (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 200 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms, or (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 200 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation
* HCC patients who were not prospective suitable or refused for any other treatment, such as surgery or local ablation therapy, or recurrent or residual tumor after other treatments.
* without evidence of extrahepatic metastasis
* All target tumors must be encompassable within single irradiation field (15x15 cm maximum)
* no previous treatment to target tumors by other forms of RT
* liver function of Child-Pugh class A or B7 (Child-Pugh score of ≤7)
* Age of ≥18 years
* performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* WBC count ≥ 2,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 25,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit of normal; no ascites)
* no serious comorbidities other than liver cirrhosis
* written informed consent

Exclusion Criteria:

* evidence of extrahepatic metastasis
* age < 18 years
* liver function of Child-Pugh class B8-9 and C (Child-Pugh score of >7)
* previous history of other forms of RT adjacent to target tumors
* poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* multicentric HCCs, except for those with the following two conditions: *multinodular aggregating HCC that could be encompassed by single clinical target volume and within single irradiation field (15x15 cm maximum) *lesions other than targeted tumor that were judged as controlled with prior surgery and/or local ablation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-06-07; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
local progression-free survival | Up to 1 year
  To evaluate the local progression-free survival (LPFS) in HCC patients treated with hypofractionated proton beam radiotherapy.

SECONDARY OUTCOMES:
overall survival | Up to 2years until study closed
  * To evaluate compliance of proton beam radiotherapy for HCC by analyzing acute and late treatment-related toxicity, such as radiation-induced hepatic toxicity and gastrointestinal tract toxicity
  * To evaluate the impact of hypofractionated proton beam radiotherapy for HCC by analyzing the tumor response rate, local disease-free survival (DFS) and overall survival (OS) rate

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hyun Kim, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided